CLINICAL TRIAL: NCT02656004
Title: Essential Oil of Eucalyptus Effect on Cardiovascular Responses During Recovery of Elderly and Isometric Resistance Exercise
Brief Title: Essential Oil of Eucalyptus Effect on Cardiovascular Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do vale do São Francisco (Other)
Responsible Party: Principal Investigator, Alfredo Anderson Teixeira de Araujo, Principal Investigator, Universidade Federal do vale do São Francisco
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: UFSaoFrancisco2
Record Dates: First submitted 2016-01-11; First posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension
Keywords: Eucalyptus; Autonomic nervous system; Isometric resistance exercise
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Essential Eucalyptus Oil (Experimental): Using a disposable face mask was inhale for ten minutes 0.25 ml of essential oil of eucalyptus measured through adjustable Pipettor 100/1000μl. Inhalation of the substance occurred immediately after the 20 minute rest period in the session Essential Oil of Eucalyptus.
  Interventions: Other: Essential Eucalyptus Oil
- Control (Experimental): In the control session the procedure was the same. Using a disposable face mask was inhale for ten minutes fresh air. Inhalation of the fresh air occurred immediately after the 20 minute rest period in the session Control.
  Interventions: Other: Control Session

INTERVENTIONS:
Other: Essential Eucalyptus Oil — Using a disposable face mask was inhale for ten minutes 0.25 ml of essential oil of eucalyptus measured through adjustable Pipettor 100/1000μl. Inhalation of the substance occurred immediately after the 20 minute rest period in the session Essential Oil of Eucalyptus.
  Arms: Essential Eucalyptus Oil
Other: Control Session — In the control session the procedure was the same. Using a disposable face mask was inhale for ten minutes fresh air. Inhalation of the fresh air occurred immediately after the 20 minute rest period in the session Control.
  Arms: Control

SUMMARY:
The essential eucalyptus oil has therapeutic potential in the cardiovascular system, with possibilities of acting on the autonomic tonus and reduction of cardiovascular overload. Hemodynamic conditions can change during the physical requirement and offer a framework of increased cardiovascular risk, especially for elderly individuals. In this sense, preservation strategies of cardiovascular autonomic control and demand in this population in conditions of rest and/or exercise are required. The aim of this study was investigate the effect of the essential eucalyptus oil on cardiovascular responses and recovery during submaximal isometric resisted exercise series in the elderly. Twenty elderly male (69.1 ± 5.7 years; 75.3 ± 12.3 kg; 168.0 ± 6.0 cm) participated in this study. Were excluded from the sample the volunteers who presented some serious illness known according to the criteria of risk stratification of the American College of Sports Medicine. In random order crusade, the volunteers were subjected to: 1) trial session through the essential eucalyptus oil and inhalation; 2) session control without inhalation of essential eucalyptus oil. After the sessions 1 and 2, the volunteers remained in recovery for a period of 60 minutes, in temperature-controlled environment and comfortably seated. After this period were performed 3 sets of isometric resisted exercise on dominant upper limb in intensity of 30% of maximum voluntary contraction in 1 min each, with 1 min recovery interval. Measures of heart rate, blood pressure, rate product pressure and heart rate variability were held in the rest for 20 min, in recovery during 60 min and during the 3 sets of isometric resisted exercise. Indicators of heart rate variability were analysed from the time and the frequency domain. ANOVA two-way for repeated measurements with Post Hoc of Tukey were employed (p<0.05).

DETAILED DESCRIPTION:
The volunteers performed in random order two experimental sessions separated by 48 hours and being: 1) Control and; 2) Inhalation Essential Oil of Eucalyptus. The experimental sessions were always performed in the morning and in the same time of day for the same volunteer, avoiding possible influences circadian rhythm. The experimental sessions were held at the Exercise Physiology Laboratory at the Federal University of Vale do São Francisco with controlled temperature 25°C. At times the pre session (rest), recovery and during the isometric resistance exercise (post-session) in upper limb by hand grip, blood pressure measurements were taken, heart rate and records of the intervals R-R in the absolute time and frequency domain, and are calculated the rate product pressure values (systolic blood pressure x heart rate). Using a disposable face mask participants inhale for ten minutes 0.25 ml of essential oil of eucalyptus measured through adjustable Pipettor 100/1000μl. Inhalation of the substance occurred immediately after the 20 minute rest period in the session Essential Oil of Eucalyptus. In the control session the volunteers remained in a similar manner, with the installed face mask, however inhaling fresh air. The test for determining the maximal voluntary contraction was held in hand grip device Hydraulic Hand Dynamometer Saehan Model SH5001 ranging from 0-90 kgf of grip and precision of 2 kgf. Before the test was performed familiarization session with two series each of 10 seconds with the minimum load allowed by the equipment, the series being separated by a 2-minute recovery period. The value of the maximum voluntary load was determined by the highest value obtained in three attempts of 10 seconds each, with 2 minutes between each trial and the position of the grip handle has been self selected. The experimental isometric resistance exercise sessions were undertaken after 48 hours of interval maximum voluntary contraction test, and the same equipment previously used for the test. The isometric resistance exercise series were held with volunteers sitting positioned comfortably and with the shoulder adducted, the elbow flexed at 90° and the forearm in neutral position, and the position of the self selected grip handle. The highest value obtained in kgf in maximum voluntary contraction test was used as a reference to calculate the absolute intensity of the exercise, which was corresponding to the relative intensity of 30% of the test. Three sets were performed with duration of 1 minute recovery at the same time in both sessions (Eucalyptus Essential Oil and Control).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and hypertensive
* Between 60 and 80 years old

Exclusion Criteria:

* Diabetic
* Morbid obesity
* Abnormality on the electrocardiogram at rest with ischemic heart suggested
* Heart disease
* Uncontrolled hypertension
* Chronic renal failure

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure response to Inhalation of Essential Eucalyptus Oil | 2 hours

IPD SHARING:
Plan to Share IPD: No